CLINICAL TRIAL: NCT05121246
Title: A Randomized, Double-Blind, 3-arm Parallel Study to Compare PK, Safety, IMM and Tolerability of MB05, EU-sourced Synagis® and US-sourced Synagis®, as a Single Dose Intramuscular Injection in Healthy Volunteers.
Brief Title: A PK Study Comparing MB05, EU-sourced Synagis® and US-sourced Synagis® in Healthy Volunteers.
Acronym: FANTASY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MB05-A-01-21
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MB05 (Proposed palivizumab biosimilar) (Experimental): Sterile vial 100mg/1ml, single-dose 3mg/kg administered as intramuscular injection on day 1.
  Interventions: Drug: MB05 (Proposed palivizumab biosimilar)
- EU-Synagis® (Active Comparator): Sterile vial 100mg/1ml, single-dose 3mg/kg administered as intramuscular injection on day 1
  Interventions: Drug: EU-Synagis®
- US-Synagis® (Active Comparator): Sterile vial 100mg/1ml, single-dose 3mg/kg administered as intramuscular injection on day 1
  Interventions: Drug: US-Synagis®

INTERVENTIONS:
Drug: MB05 (Proposed palivizumab biosimilar) — Single IM dose of 3 mg/kg
  Arms: MB05 (Proposed palivizumab biosimilar)
Drug: EU-Synagis® — Single IM dose of 3 mg/kg
  Arms: EU-Synagis®
Drug: US-Synagis® — Single IM dose of 3 mg/kg
  Arms: US-Synagis®

SUMMARY:
During the course of the study, the similarity in pharmacokinetics will be assessed by sampling the levels of drug in the blood, and by comparing these levels among the different administration arms. Safety, tolerability, and immunologic response to the administered drugs will also be evaluated throughout.

DETAILED DESCRIPTION:
MB05 is being developed as a potential biosimilar to Synagis® for all indications for which Synagis® is approved. This study is designed to demonstrate PK similarity of the proposed biosimilar test product MB05 and the reference products EU- and US-Synagis®.This is a first-in-human study of the Synagis® biosimilar MB05. The reference product ynagis® was first approved by the US Food and Drug Administration (FDA) in 1998 and by the European Medicines agency (EMA) in 1999.

As a proposed biosimilar, the clinical experience with Synagis® (as described in the Synagis® summary of product characteristics) (most recent versions) is deemed applicable to MB05.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers will be included in the study if they meet all of the following criteria at screening, and after check-in on Day -1 (prior to dose administration on Day 1):

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adult male and female volunteers, 18 to 55 years of age (inclusive).
3. Body mass index (calculated) within the range of 18 to 30 kg/m2 inclusive and total body weight between 50 and 95 kg, inclusive, at screening and check-in.
4. Medically healthy without clinically significant abnormalities, including:

   1. Physical examination without any clinically significant findings, in the opinion of the Investigator.
   2. Systolic blood pressure (BP) in the range of 90 to 145 mm Hg (inclusive) and diastolic BP in the range of 50 to 90 mm Hg (inclusive) after at least 5 minutes in the supine position.
   3. Pulse rate (PR) in the range of 40 to 100 beats/min (inclusive) after at least 5 minutes rest in a supine position.
   4. Normal body temperature 35.1 to 37.6°C (inclusive) (Tympanic temperature).
   5. Triplicate 12-lead electrocardiogram (ECG), taken after the volunteer has been supine for at least 5 minutes, with a QT interval corrected using the Fridericia method (QTcF) ≤ 450 msec for males and ≤ 470 msec for females and no clinically significant abnormalities, in the opinion of the Investigator.
   6. Adequate bone marrow function defined by absolute neutrophil count, platelet count and haemoglobin levels within normal ranges (per local laboratory standard).
   7. Adequate liver function as defined by:

      • Alanine aminotransferase (ALT) aspartate aminotransferase (AST), alkaline phosphatase (ALP) and bilirubin ≤ 1.5 x upper limit of normal (ULN). Note: Bilirubin > 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is < 35%.
   8. Adequate coagulation, as defined by:

      • Prothrombin time (PT) / International Normalised Ratio (INR), thrombin time (TT), or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN.
   9. Adequate renal function, as defined by:

      • Creatinine or measured or calculated creatinine clearance ≤ 1.5 x ULN. Note. Glomerular filtration rate (GFR) can be used in place of creatinine or CrCl.
   10. No other clinically significant findings in serum chemistry, haematology, coagulation and urinalysis examinations, in the opinion of the Investigator.

   Note. The above assessments may be repeated once, if abnormal values were recorded in the first instance, at the discretion of the Investigator.
5. No prior history of chronic alcohol abuse or excessive alcohol intake, at the discretion of the PI, within 12 weeks prior to screening, and negative alcohol test results (at screening and on Day -1). Excessive alcohol intake is defined as regular consumption of > 12 standard units of alcohol per week, or more than 4 standard drinks on > 3 days per week, where 1 standard drink is 10 g of pure alcohol and is equivalent to 285 mL beer [4.9% Alc./Vol], 100 mL wine [12% Alc./Vol], 30 mL spirit [40% Alc./Vol]).
6. No prior history of substance abuse or drug addiction within 12 months prior to first study drug administration and negative drug test results (at screening and on Day -1).
7. Female volunteers must:

   1. Be of non-childbearing potential i.e., surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before the Screening visit) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle-stimulating hormone [FSH] level indicative of postmenopausal status per local laboratory definition), OR
   2. If of childbearing potential:

      * Must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test within 24 hours prior to dose administration on Day 1
      * Must not be breastfeeding, lactating or planning pregnancy during the study period
      * Must agree not to attempt to become pregnant
      * If not exclusively in same-sex relationships, must agree to use adequate contraception (which is defined as use of a condom by the male partner combined with the use of a highly effective method of contraception per APPENDIX 4) from 30 days prior to dosing until at least 190 days after the last dose of study drug.
      * Must agree not to donate ova for at least 190 days after the last dose of study drug.
8. Male volunteers, must agree not to donate sperm for at least 190 days after the last dose of study drug, and if engaging in sexual intercourse, must agree to:

   1. use a condom, PLUS
   2. when engaging in sexual intercourse with a female who may become pregnant, must agree to have the female use an acceptable form of contraception (refer to APPENDIX 4) from 30 days prior to dosing until at least 190 days after the last dose of study drug.
9. Have suitable venous access for blood sampling.
10. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

Healthy volunteers will be excluded from the study if there is evidence of any of the following at screening or any time after check-in on Day -1 (prior to dose administration on Day 1):

1. Prior exposure to Synagis® (palivizumab).
2. Have a history of hypersensitivity or allergic reactions (either spontaneous or following drug administration) to any drug compound or its excipients, food, or other substance. Minor (non-anaphylactic) reactions to food substances (non-excipients) may be permitted, at the discretion of the Investigator.
3. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, deemed to be clinically relevant as determined by the Investigator (or designee).
4. Presence or evidence of recent sunburn, scar tissue, tattoo (more than 25% of body area), open sore or branding that, in the opinion of the Investigator, would interfere with interpretation of skin adverse reactions.
5. Have a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) or human immunodeficiency virus (HIV). Screening only.
6. Have a positive test result for COVID-19 (polymerase chain reaction [PCR] or antigen test) within 72 hours prior to dose administration.
7. If subject smokes, subject is unwilling to abstain from smoking for 7 days prior to admission and during the confinement period.
8. Positive serum pregnancy test for women of childbearing potential (WOCBP) at the screening visit or positive urine pregnancy test with confirmatory serum pregnancy test prior to dosing on Day 1.
9. Females who are breastfeeding.
10. Have a history of cancer including lymphoma, leukaemia and skin cancer (volunteers with surgically resected basal cell carcinoma or squamous cell carcinomas are permitted).
11. Have an illness within 30 days prior to screening, or prior to dosing, that is classed as clinically significant by the Investigator.
12. Any clinically significant infection, in the opinion of the Investigator, ongoing at screening or admission to the clinical unit.
13. Prior exposure to any investigational monoclonal antibody within 6 months or 5 half-lives of the previous drug (if known), whichever is longer, prior to study drug administration.
14. Have been dosed in another clinical study with an investigational drug (excluding monoclonal antibody) within 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to the administration of the study drug or are currently participating in another clinical study of an investigational drug or intending to participate in another clinical study of an investigational drug before completion of all scheduled evaluations in this clinical study.
15. Have had major surgery within 30 days prior to screening or will have an operation between screening and the end of study visit.
16. Have donated > 100 mL blood or plasma within 4 weeks prior to the administration of the study drug. Participant must also agree to refrain from donating blood or blood products throughout the duration of the study.
17. Use of any prescription or over-the-counter medication (including herbal products, diet aids, and hormone supplements) within 10 days or 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, which, in the opinion of the Investigator, could affect the outcome of the study. The following exceptions apply:

    1. Contraceptives for WOCBP.
    2. Paracetamol (up to a maximum of 4 doses of 500 mg per day, and no more than 3g per week).
    3. Ibuprofen (up to a maximum of 4 doses of 200 mg per day).
18. Has received (or plans to receive) a vaccine within the following timeframes:

    1. Live or attenuated vaccine within 3 months prior to dose administration on Day 1 or plans to receive a live or live attenuated vaccine during the study.
    2. Other vaccines (including COVID-19 vaccines) within 14 days prior to dose administration on Day 1 or plans to receive other vaccines within 14 days following dose administration on Day 1.
19. Any person who is an employee of an Investigator or Sponsor, or an immediate relative of an Investigator.
20. Any other condition or prior therapy that in the opinion of the Investigator would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Nucleus Network. Q-Pharm Pty Ltd, Brisbane, Queensland, Australia
- New Zealand (2):
  - New Zealand Clinical Research Ltd., Auckland
  - New Zealand Clinical Research Ltd., Christchurch

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 150 subjects were enrolled into the study, of those, 9 subjects were randomized but not dosed for reasons outlined as follows:
  * Five subjects were unable to be dosed due to dosing delays at the site. These subjects were discharged from the clinical unit as eligible;
  * One subject was not dosed due a randomization error;
  * One subject did not meet inclusion criterion #9 ;
  * Two subjects did not meet inclusion criteria #4
Groups:
- Arm A: 3 mg/kg MB05
- Arm B: 3 mg/kg EU-Synagis®
- Arm C: 3 mg/kg US-Synagis®
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 46 | 48 | 47
Completed | 46 | 47 | 44
Not Completed | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Of 150 subjects enrolled, a total of 9 subjects were randomized but did not receive a dose of IP, for reasons outlined as follows:
  * Five subjects were unable to be dosed due to dosing delays at the site. These subjects were discharged from the clinical unit as eligible;
  * One subject was not dosed due a randomization error;
  * One subject did not meet inclusion criterion #9;
  * Two subjects did not meet inclusion criteria #4
Groups:
- Total: Total of all reporting groups
Arm/Group | MB05 (Proposed Palivizumab Biosimilar) | EU-Synagis® | US-Synagis® | Total
Number analyzed (Participants) | 46 | 48 | 47 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 46 | 48 | 47 | 141
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (8.9) | 31.8 (10.6) | 30.4 (9.4) | 31.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 31 | 27 | 83
  Male | 21 | 17 | 20 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6 | 12
  Not Hispanic or Latino | 40 | 43 | 38 | 121
  Unknown or Not Reported | 2 | 3 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 6 | 9 | 8 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 4 | 6
  Black or African American | 0 | 0 | 1 | 1
  White | 37 | 36 | 31 | 104
  More than one race | 0 | 1 | 2 | 3
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Pharmacokinetic (PK) Profiles Between MB05 and EU-Synagis®, Between MB05 and US-Synagis® and Between EU-Synagis® and US-Synagis® in Terms of Area Under the Serum Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf)
Description: Bioequivalence between MB05 and EU Synagis®, between MB05 and US-Synagis® and between EU-Synagis® and US-Synagis® will be investigated for AUC0-inf and Cmax by analysis of variance using log-transformed PK parameter values. Bioequivalence will be assessed by calculating the 90% CIs for the ratio of the least squares geometric means for each pairwise comparison and each PK parameter. Bioequivalence will be concluded where the 90% CIs for the ratio of least squares geometric means are contained within the range 80.00% to 125.00%.
  Blood samples collection timepoints: pre-dose (within 60 minutes prior); 4 hr (+/- 15 min); 12 hr (+/- 15 min); 24 hr (+/- 1 hr); 48 hr (+/- 5 hr); 72 hr (+/- 5 hr); 96 hr (+/- 5 hr); 120 hr (+/- 5 hr); 168 hr (+/- 5 hr) post-dose, and then at Days 15; 22; 29; 36; 43; 57; 71; 85; and 99 (end of study).
Time Frame: Day 1 - Day 100
Population: The PK population will include all randomized participants where there is sufficient data for reliable estimates of AUC0-inf (as determined by the study Pharmacokineticist).
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Groups:
- MB05 vs EU-Synagis®: 3 mg/kg MB05 proposed palivizumab biosimilar /3 mg/kg EU-Synagis®
- MB05 vs US-Synagis®: 3 mg/kg MB05 /3 mg/kg US-Synagis®
- EU-Synagis® vs US-Synagis®: 3 mg/kg EU-Synagis® /3 mg/kg US-Synagis®
Arm/Group | MB05 vs EU-Synagis® | MB05 vs US-Synagis® | EU-Synagis® vs US-Synagis®
Number analyzed (Participants) | 94 | 93 | 95
ratio | 104.9 [86.9 to 126.6] | 101.1 [84.6 to 120.7] | 96.3 [81.3 to 114.2]
Statistical Analysis 1: Comparison: MB05 vs EU-Synagis® vs MB05 vs US-Synagis® vs EU-Synagis® vs US-Synagis®; PK parameters will be determined using a non-compartmental analysis method. Bioequivalence between MB05 and EU-Synagis®, between MB05 and US-Synagis® and between EU-Synagis® and US-Synagis® will be established by analysis of variance for the PK parameters AUC0-inf, and Cmax; Test type: Equivalence — CI 90% of least squares geometric means must be entirely contained within the range [80%-125%]; PK parameters for each participant will be listed and summarised by treatment using descriptive statistics

2. Primary Outcome: Compare the Pharmacokinetic (PK) Profiles Between MB05 and EU-Synagis®, Between MB05 and US-Synagis® and Between EU-Synagis® and US-Synagis® in Terms of Maximum Observed Serum Concentration Cmax.
Description: as for outcome 1
Time Frame: Day 1 - Day 100
Population: The PK population will include all randomized participants where there is sufficient data for reliable estimates of Cmax (as determined by the study Pharmacokineticist).
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | MB05 vs EU-Synagis® | MB05 vs US-Synagis® | EU-Synagis® vs US-Synagis®
Number analyzed (Participants) | 94 | 93 | 95
ratio | 100.4 [80.2 to 125.8] | 96.9 [79.7 to 117.8] | 96.5 [78.4 to 118.6]
Statistical Analysis 1: Comparison: MB05 vs EU-Synagis® vs MB05 vs US-Synagis® vs EU-Synagis® vs US-Synagis®; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — CI 90% of least squares geometric means must be entirely contained within the range [80%-125%]; PK parameters for each participant will be listed and summarised by treatment using descriptive statistics

3. Primary Outcome: Pharmacokinetics (PK)- (AUC0-inf)
Description: Pharmacokinetic (PK) profiles for each arm (AUC0-inf)
Time Frame: Day 1 - Day 100
Population: The PK population included all randomized participants where there was sufficient data for reliable estimates of Cmax (as determined by the study Pharmacokineticist). Participants with dosing or PK sampling deviations that could potentially affect the PK profile were also excluded from the PK population, at the discretion of the study Pharmacokineticist. The PK population was used for the summaries of all PK data.
Measure: Mean (Standard Error); unit: h*µg/mL
Arm/Group | MB05 (Proposed Palivizumab Biosimilar) | EU-Synagis® | US-Synagis®
Number analyzed (Participants) | 46 | 48 | 47
h*µg/mL | 20100 (45.0) | 19100 (48.9) | 19300 (44.0)

4. Primary Outcome: Pharmacokinetics (PK) - (Cmax)
Description: Pharmacokinetic (PK) profiles for each arm (Cmax)
Time Frame: Day 1 - Day 100
Population: The PKS included all randomized subjects who received any amount of study treatment and where there was sufficient data for reliable estimates of Cmax (as determined by the study Pharmacokineticist). The PKS was used for the summaries of all PK data. All 141 subjects in the SS had sufficient samples collected to construct an evaluable concentration-time profile, and so were included in PK analysis set.
Measure: Mean (Standard Error); unit: µg/mL
Arm/Group | MB05 (Proposed Palivizumab Biosimilar) | EU-Synagis® | US-Synagis®
Number analyzed (Participants) | 46 | 48 | 47
µg/mL | 22.5 (57.0) | 22.7 (56.1) | 22.2 (53.4)

5. Secondary Outcome: Tmax
Description: Time to reach maximum observed serum concentration (Cmax)
Time Frame: Day 1 - Day 100
Measure: Median (90% Confidence Interval); unit: h
Groups:
- MB05 (Proposed Palivizumab Biosimilar): 3 mg/kg MB05 proposed palivizumab biosimilar
- EU-Synagis®: 3 mg/kg EU-Synagis®
- US-Synagis®: 3 mg/kg US-Synagis®
Arm/Group | MB05 (Proposed Palivizumab Biosimilar) | EU-Synagis® | US-Synagis®
Number analyzed (Participants) | 46 | 48 | 47
h | 124 [48.0 to 506] | 120 [46.4 to 360] | 124 [46.6 to 528]

6. Secondary Outcome: t1/2
Description: Apparent terminal elimination half-life (t1/2)
Time Frame: Day 1 - Day 100
Measure: Mean (Standard Error); unit: h
Arm/Group | MB05 (Proposed Palivizumab Biosimilar) | EU-Synagis® | US-Synagis®
Number analyzed (Participants) | 46 | 48 | 47
h | 586 (26.6) | 562 (27.9) | 559 (30.8)

7. Secondary Outcome: Vz
Description: Apparent volume of distribution (Vz)
Time Frame: Day 1- Day 100
Measure: Mean (Standard Error); unit: mL
Arm/Group | MB05 (Proposed Palivizumab Biosimilar) | EU-Synagis® | US-Synagis®
Number analyzed (Participants) | 46 | 48 | 47
mL | 11500 (63.7) | 11400 (66.5) | 9400 (37.3)

8. Secondary Outcome: CL
Description: Apparent total serum clearance ((CL)
Time Frame: Day 1- Day 100
Measure: Mean (Standard Error); unit: mL/h
Arm/Group | MB05 (Proposed Palivizumab Biosimilar) | EU-Synagis® | US-Synagis®
Number analyzed (Participants) | 46 | 48 | 47
mL/h | 14.8 (80.7) | 14.6 (66.3) | 12.8 (49.9)

9. Secondary Outcome: Safety and Tolerability
Description: Treatment-related Adverse Events
Time Frame: Day 1- Day 100
Population: The safety population will include all randomized participants who received any amount of study treatment and will be summarized according to the treatment actually received, if this differs from that to which the participant was randomized to. The safety population will be used for the summaries of all safety, baseline and demographic data.
Measure: Number; unit: participants
Arm/Group | MB05 (Proposed Palivizumab Biosimilar) | EU-Synagis® | US-Synagis®
Number analyzed (Participants) | 46 | 48 | 47
participants
  Any TEAE | 33 | 36 | 29
  Any Treatment-Related TEAE | 7 | 14 | 6
  Any Serious TEAE | 0 | 0 | 0
  Any TEAE that is an injection site reaction | 5 | 15 | 6
  Any TEAE leading to death | 0 | 0 | 0
  Any TEAE leading to study withdrawal | 0 | 0 | 0

10. Secondary Outcome: Immunogenicity
Description: Assessment of anti-drug antibodies (ADA) against palivizumab
Time Frame: Day 1- Day 100
Population: The immunogenicity population will include all randomized participants who receive any amount of study treatment and who have at least 1 evaluable immunogenicity parameter post-dose and will be summarized according to the treatment actually received, if this differs from that to which the participant was randomized. The immunogenicity population will be used for the summaries of all immunogenicity data.
Measure: Number; unit: participants
Arm/Group | MB05 (Proposed Palivizumab Biosimilar) | EU-Synagis® | US-Synagis®
Number analyzed (Participants) | 46 | 48 | 47
participants
  Baseline ADA positive | 3 | 1 | 3
  Baseline ADA negative | 43 | 47 | 44
  Treatment-induced ADA positive | 29 | 40 | 28
  Treatment-boosted ADA positive | 1 | 1 | 2
  ADA negative | 16 | 7 | 17

ADVERSE EVENTS:
Time Frame: Day 1 to Day 100
Description: For all AEs reported, the actions taken and outcomes must be specified and documented in the eCRF and appropriate form(s) (where required) as described in the eCRF completion guidelines.
Arm/Group | MB05 (Proposed Palivizumab Biosimilar) | EU-Synagis® | US-Synagis®
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 0/46 | 0/48 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT05121246/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT05121246/SAP_001.pdf